CLINICAL TRIAL: NCT04936438
Title: Clinical Cohort Study - INTERCATH: A Diseased Cohort Based Epidemiologic, Prospective, Single Center Cohort Study for Novel Research in Cardiovascular Risk Prediction Using a Sophisticated Biobank
Brief Title: Clinical Cohort Study - INTERCATH
Status: Active, not recruiting | Type: Observational
Sponsor: University of Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Fabian J Brunner, MD, Co-principal investigator, University of Hamburg-Eppendorf
Other Study IDs: INTERCATH
Record Dates: First submitted 2021-06-12; First posted 2021-06-23 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Coronary Artery Disease; Coronary Disease; Coronary Syndrome; SCAD; Cardiovascular Diseases
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Angina, Unstable; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Within a CAD patient cohort there is a wide variability of clinical manifestation and severity of coronary disease. Distinct determinants that would explain the variety of CAD phenotypes with differing prognosis are yet undiscovered. Aim of this study is to find genetic variants, biomarkers, and clinical cardiovascular risk factors that relate to specific coronary artery disease phenotypes and related pathologies in a patient population.

DETAILED DESCRIPTION:
Atherosclerotic Coronary Artery Disease (CAD) is one of the leading causes of death in industrialized countries and accounts for a high lifetime prevalence. Within a CAD patient cohort there is a broad inter-individual difference with regard to clinical manifestation and severity of disease, e.g. stable angina vs. acute coronary syndrome, calcified vs. thrombotic coronary lesions or one vessel vs. complex three vessel disease or left main stenosis. Thus, depending on the CAD phenotype there is a broad difference in CAD patients' prognosis. Similarly, other non-atherosclerotic coronary pathologies such as Spontaneous Coronary Dissection (SCAD) are related with devastating illness in mainly young patients. For these patients there is an unmet need in the knowledge of epidemiology, presentation, current management and outcome. Aim of this study is to discover genetic variants, biomarkers, and clinical cardiovascular risk factors that relate to specific CAD (and related coronary pathologies) phenotypes in a national patient population. This may allow an improvement of individualized risk stratification and contribute to discover pathways in the pathogenesis and open the avenue for potential therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a minimum age of 18 years
* Any patient with an available complete coronary angiography
* Ability to provide written informed consent in accordance with Good Epidemiological Practice and local legislation

Exclusion Criteria:

* Physical or psychological incapability to take part in the study
* Known anaemia (Hemoglobin < 7.5 g/dl)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient undergoing coronary angiography.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with non-fatal or fatal major adverse cardiovascular events (MACE) | Through study completion, an average of 5 years
  MACE as a composite endpoint consists of
  * occurrence of non-fatal and fatal myocardial infarction
  * occurrence of non-fatal and fatal stroke
  * need for coronary revascularization (percutaneous coronary intervention or coronary bypass graft operation)
  Endpoints will be recorded by telephone interview during census follow up. All endpoint information will be validated by official medical records.
All-cause mortality | Through study completion, an average of 5 years
  Information from the population register will be used to assess all-cause mortality.

CONTACTS AND LOCATIONS:
Locations (1):
- University Heart and Vascular Center Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Blaum C, Seiffert M, Gossling A, Kroger F, Bay B, Lorenz T, Braetz J, Graef A, Zeller T, Schnabel R, Clemmensen P, Westermann D, Blankenberg S, Brunner FJ, Waldeyer C. The need for PCSK9 inhibitors and associated treatment costs according to the 2019 ESC dyslipidaemia guidelines vs. the risk-based allocation algorithm of the 2017 ESC consensus statement: a simulation study in a contemporary CAD cohort. Eur J Prev Cardiol. 2021 Mar 23;28(1):47-56. doi: 10.1093/eurjpc/zwaa088. PMID 33580772
- [Result] Brunner FJ, Kroger F, Blaum C, Gossling A, Lorenz T, van Erckelens E, Bratz J, Westermann D, Blankenberg S, Zeller T, Waldeyer C, Seiffert M. Association of high-sensitivity troponin T and I with the severity of stable coronary artery disease in patients with chronic kidney disease. Atherosclerosis. 2020 Nov;313:81-87. doi: 10.1016/j.atherosclerosis.2020.09.024. Epub 2020 Sep 28. PMID 33032237
- [Result] Blaum C, Brunner FJ, Kroger F, Braetz J, Lorenz T, Gossling A, Ojeda F, Koester L, Karakas M, Zeller T, Westermann D, Schnabel R, Blankenberg S, Seiffert M, Waldeyer C. Modifiable lifestyle risk factors and C-reactive protein in patients with coronary artery disease: Implications for an anti-inflammatory treatment target population. Eur J Prev Cardiol. 2021 Apr 10;28(2):152-158. doi: 10.1177/2047487319885458. Epub 2019 Nov 10. PMID 33838040
- [Result] Waldeyer C, Brunner FJ, Braetz J, Ruebsamen N, Zyriax BC, Blaum C, Kroeger F, Kohsiack R, Schrage B, Sinning C, Becher PM, Karakas M, Zeller T, Westermann D, Sydow K, Blankenberg S, Seiffert M, Schnabel RB. Adherence to Mediterranean diet, high-sensitive C-reactive protein, and severity of coronary artery disease: Contemporary data from the INTERCATH cohort. Atherosclerosis. 2018 Aug;275:256-261. doi: 10.1016/j.atherosclerosis.2018.06.877. Epub 2018 Jun 22. PMID 29980052
- [Result] Waldeyer C, Seiffert M, Staebe N, Braetz J, Kohsiack R, Ojeda F, Schofer N, Karakas M, Zeller T, Sinning C, Schrage B, Westermann D, Sydow K, Blankenberg S, Brunner FJ, Schnabel RB. Lipid Management After First Diagnosis of Coronary Artery Disease: Contemporary Results From an Observational Cohort Study. Clin Ther. 2017 Nov;39(11):2311-2320.e2. doi: 10.1016/j.clinthera.2017.10.005. Epub 2017 Nov 2. PMID 29103665
- [Result] Zeller T, Seiffert M, Muller C, Scholz M, Schaffer A, Ojeda F, Drexel H, Mundlein A, Kleber ME, Marz W, Sinning C, Brunner FJ, Waldeyer C, Keller T, Saely CH, Sydow K, Thiery J, Teupser D, Blankenberg S, Schnabel R. Genome-Wide Association Analysis for Severity of Coronary Artery Disease Using the Gensini Scoring System. Front Cardiovasc Med. 2017 Sep 20;4:57. doi: 10.3389/fcvm.2017.00057. eCollection 2017. PMID 28979897
- [Derived] Bay B, Fuh MM, Rohde J, Worthmann A, Gossling A, Arnold N, Koester L, Lorenz T, Blaum C, Kirchhof P, Blankenberg S, Seiffert M, Brunner FJ, Waldeyer C, Heeren J. Sex differences in lipidomic and bile acid plasma profiles in patients with and without coronary artery disease. Lipids Health Dis. 2024 Jun 26;23(1):197. doi: 10.1186/s12944-024-02184-z. PMID 38926753
- [Derived] Bay B, Gossling A, Blaum CM, Kroeger F, Koppe L, Lorenz T, Koester L, Clemmensen P, Westermann D, Kirchhof P, Blankenberg S, Zeller T, Seiffert M, Waldeyer C, Brunner FJ. Association of High-Sensitivity Troponin T and I Blood Concentrations With All-Cause Mortality and Cardiovascular Outcome in Stable Patients-Results From the INTERCATH Cohort. J Am Heart Assoc. 2022 Sep 6;11(17):e024516. doi: 10.1161/JAHA.121.024516. Epub 2022 Jul 19. PMID 35862141